CLINICAL TRIAL: NCT03467503
Title: Healthy Diet for Healthy Moms and Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Arpita Basu, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1155039
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Gestational Diabetes; Obesity; Pregnancy, High Risk
MeSH Terms: conditions — Diabetes, Gestational; Obesity | interventions — blueberry extract

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal Care/Nutrition Education (No Intervention): Participants were given nutrition educational counseling on healthy dietary habits and gestational weight gain as part of standard prenatal care.
- Dietary Intervention (Experimental): Participants were given dietary blueberries (2 cups) and soluble fiber (12g). They also received nutrition educational counseling on healthy dietary habits and gestational weight gain as part of standard prenatal care.
  Interventions: Dietary Supplement: Blueberry + soluble fiber

INTERVENTIONS:
Dietary Supplement: Blueberry + soluble fiber — Dietary frozen blueberries and soluble fiber for 20 weeks
  Arms: Dietary Intervention

SUMMARY:
The purpose of this clinical study is to collect baseline information on dietary habits and metabolic risk factors, and to examine the effects of a dietary intervention focusing on fiber and antioxidant rich berries on the development of gestational diabetes, maternal glucose and lipid control and inflammation in obese pregnant women at risk of developing diabetes. With the ongoing epidemic of obesity, the prevalence of gestational diabetes is significantly increasing and the goal of this research is to identify optimal dietary strategies that can reverse this condition or control the rise in blood glucose among those with already developed diabetes.

ELIGIBILITY:
Inclusion Criteria:

* BMI > or = 30, <20 weeks gestation and singleton pregnancy with the following options: previous history of gestational diabetes and/or family history of diabetes

Exclusion Criteria:

* • Twin or multiple pregnancy

  * Chronic pre-pregnancy conditions (CHD, cancer, diabetes)
  * Gastrointestinal conditions
  * Anemia
  * Allergic to berries and fiber
  * Vegetarian food habits or special diets
  * Not proficient in English and/or unable to provide consent

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy study
Enrollment: 34 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | 20 weeks
  Maternal weight gain in lbs
Gestational glycemia | 20 weeks
  Maternal blood glucose and HbA1c as measures of glycemia
Maternal serum lipids | 20 weeks
  Conventional total, LDL-cholesterol and their particle size to describe lipid profiles
Maternal inflammation | 20 weeks
  C-reactive protein as a stable biomarker of inflammation

SECONDARY OUTCOMES:
Maternal biomarkers of atherosclerosis | 20 weeks
  Serum cytokines measured as interleukins and adipokines
Maternal dietary intakes | 20 weeks
  Maternal intakes of energy intake and nutrients

OTHER OUTCOMES:
Maternal metabolomics | 20 weeks
  Maternal serum NMR metabolites

CONTACTS AND LOCATIONS:
Overall Officials: Arpita Basu, PhD, Principal Investigator — University of Nevada at Las Vegas
Locations (1):
- University of Nevada at Las Vegas, Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Basu A, Feng D, Planinic P, Ebersole JL, Lyons TJ, Alexander JM. Dietary Blueberry and Soluble Fiber Supplementation Reduces Risk of Gestational Diabetes in Women with Obesity in a Randomized Controlled Trial. J Nutr. 2021 May 11;151(5):1128-1138. doi: 10.1093/jn/nxaa435. PMID 33693835